CLINICAL TRIAL: NCT02809326
Title: Trauma Management Therapy for OEF and OIF Combat Veterans
Acronym: TMT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Central Florida (Other)
Responsible Party: Principal Investigator, Deborah Beidel, Pegasus Professor of Psychology and Medical Education Associate Chair for Research Director, UCF RESTORES, University of Central Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UCFlorida
Record Dates: First submitted 2016-05-10; First posted 2016-06-22 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Post-Traumatic Stress Disorder; Combat Disorders
Keywords: efficiency; exposure therapy; PTSD; combat; veterans
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Combat Disorders | interventions — Implosive Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 17 week Trauma Management Therapy (TMT) (Experimental): TMTconsists of 29 treatment sessions administered over a period of 3 weeks. Individual VR-assisted exposure sessions (14 sessions) are followed by Social and Emotional Regulation (SER) sessions conducted in small groups. Individual exposure therapy includes virtual reality to assist in augmenting exposure therapy. Group therapy includes anger management, social skills training, problem solving and behavioral activation for depression. The treatment program as a whole results in approximately 43.5 hours of therapist contact for each patient.
  Interventions: Behavioral: Trauma Management Therapy
- 3 week Trauma Management Therapy (TMT) (Experimental): Intensive 3-Week Trauma Management Therapy consists of 29 treatment sessions administered over a period of 3 weeks. Individual VR-assisted exposure sessions and group sessions are conducted Monday-Friday with individual sessions conducted in the morning and Social and Emotional Regulation (SER) sessions conducted in the afternoon. Education and exposure are implemented individually while SER is administered in small group sessions (3-5 people). All exposure treatment sessions will terminate after a decline of 50% in the highest rating recorded. SER sessions will be 90 minutes. The treatment program as a whole results in approximately 43.5 hours of therapist contact for each patient.
  Interventions: Behavioral: Intensive 3-Week Trauma Management Therapy
- 17 week Exposure Therapy Control Arm (Active Comparator): The Control Arm of the study contains 15 individual VR-assisted exposure therapy sessions and 14 psychoeducational group sessions conducted over a period of 17 weeks. After the Education session, treatment occurs three times a week during the Virtual Reality (VR) assisted Exposure phase, and then once a week during the Psychoeducational phase.The psychoeducational group therapy, will include topics such as: DSM-IV criteria of PTSD, prevalence of PTSD, risk factors for PTSD, biological and conditioning models of PTSD, PTSD comorbidity, pharmacological treatment of PTSD, the impact of substance abuse, impairment in interpersonal functioning among veterans with PTSD, and issues related to anger control problems and suggested coping strategies
  Interventions: Behavioral: 17 week Exposure Therapy Control Arm

INTERVENTIONS:
Behavioral: 17 week Exposure Therapy Control Arm — 15 individual VR-assisted exposure therapy sessions and 14 psychoeducational group sessions conducted over a period of 17 weeks. After the Education session, treatment occurs three times a week during the Virtual Reality (VR) assisted Exposure phase, and then once a week during the Psychoeducational phase.The psychoeducational group therapy, will include topics such as: DSM-IV criteria of PTSD, prevalence of PTSD, risk factors for PTSD, biological and conditioning models of PTSD, PTSD comorbidity, pharmacological treatment of PTSD, the impact of substance abuse, impairment in interpersonal functioning among veterans with PTSD, and issues related to anger control problems and suggested coping strategies
  Other Names: Exposure Therapy, Psychoeducation
  Arms: 17 week Exposure Therapy Control Arm
Behavioral: Trauma Management Therapy — TMT consists of 29 treatment sessions administered over a period of 17 weeks. After the Education session, treatment occurs three times a week during the Virtual Reality (VR) assisted Exposure phase, and then once a week during Social and Emotional Regulation (SER). Education and exposure are implemented individually while SER is administered in small group sessions (3-5 people). All exposure treatment sessions will terminate after a decline of 50% in the highest rating recorded. SER sessions will be 90 minutes. The treatment program as a whole results in approximately 43.5 hours of therapist contact for each patient.
  Other Names: TMT
  Arms: 17 week Trauma Management Therapy (TMT)
Behavioral: Intensive 3-Week Trauma Management Therapy — Intensive 3-Week Trauma Management Therapy consists of 29 treatment sessions administered over a period of 3 weeks. Individual VR-assisted exposure sessions and group sessions are conducted Monday-Friday with individual sessions conducted in the morning and Social and Emotional Regulation (SER) sessions conducted in the afternoon. Education and exposure are implemented individually while SER is administered in small group sessions (3-5 people). All exposure treatment sessions will terminate after a decline of 50% in the highest rating recorded. SER sessions will be 90 minutes. The treatment program as a whole results in approximately 43.5 hours of therapist contact for each patient.
  Other Names: Intensive TMT
  Arms: 3 week Trauma Management Therapy (TMT)

SUMMARY:
This trial will evaluate the efficacy and efficiency of Trauma Management Therapy (TMT; Frueh, Turner, Beidel, 1996; Beidel, Frueh, Uhde, under preparation), which combines individual virtual reality (VR) assisted exposure therapy with group social and emotional rehabilitation skills training (will be superior to a treatment consisting of the same VR- exposure and group psychoeducational group therapy. TMT will be conducted in traditional 17-week format, and a 3-week intensive treatment format. Outcome will be assessed using relevant clinical, process, and cost outcomes. Additionally, investigators will assess the potential of olfactory stimulation as a trigger for PTSD symptoms of intrusive thoughts and re-experiencing. Therefore, this proposal will integrate clinical and neurobiological assessment studies designed to understand the role of these factors in the etiology, maintenance, and treatment of PTSD.

DETAILED DESCRIPTION:
Background: Troop deployment for OIF/OEF has been extensive for the past five years Among returning veterans, up to 18.5% are diagnosed with posttraumatic stress disorder (PTSD). In addition to its positive symptoms (intrusive thoughts, reexperiencing, hyperarousal, and avoidance), PTSD is associated with social maladjustment, poor quality of life, medical comorbidity, and general symptom severity. Social and emotional problems include social avoidance, guilt, anger, and unemployment, impulsive or violent behavior, and family discord. A majority (> 90%) of veterans seeking treatment for PTSD also seek disability compensation for debilitating occupational impairment and there are virtually no administrative or research data to indicate veterans are recovering from PTSD. Exposure therapy, which operates on long-established and fundamental principles of behavior therapy, offers hope for acute symptom alleviation, but may not address severe social impairment.

Objectives/Hypothesis: To test the hypothesis that Trauma Management Therapy (TMT), which combines individual virtual reality (VR) assisted exposure therapy with group social and emotional rehabilitation skills training (will be superior to a treatment consisting of the same VR- exposure and group psychoeducational group therapy. Outcome will be assessed using relevant clinical, process, and cost outcomes. Additionally, we will assess the potential of olfactory stimulation as a trigger for PTSD symptoms of intrusive thoughts and re-experiencing. Therefore, this proposal will integrate clinical and neurobiological assessment studies designed to understand the role of these factors in the etiology, maintenance, and treatment of PTSD.

Specific Aims: There are three specific aims: First, we will evaluate the efficacy of Trauma Management Therapy (TMT) for the treatment of PTSD in OIF/OEF and determine if TMT (which combines exposure and social/emotional rehabilitation) improves social/emotional functioning compared to our comparison group (exposure plus psychoeducational group therapy). Second, we will explore olfactory activation patterns that may aid understanding of brain mechanisms in PTSD. Third, we will determine TMT's cost efficacy using treatment expenses and resource utilization measures.

Study Design: In a prospective randomized clinical trial we will test the superiority of TMT for OIF/OEF veterans with PTSD compared to exposure therapy plus psychoeducational group therapy. TMT combines VR assisted exposure therapy (VR-EXP) with social and emotional rehabilitation (SER). In addition to clinical, process, and cost outcomes relevant to PTSD for this population, we will include fMRI assessment of the central olfactory system in order to document its hypothesized role in fear acquisition and maintenance. Relevant outcome domains will be reassessed at mid-treatment, post-treatment, and 3- and 6-month follow-up.

ELIGIBILITY:
Inclusion criteria:

Veterans or active duty military personnel with combat-related PTSD as a result of deployment to Iraq or Afghanistan.

Exclusion criteria:

1. Personnel with acute cardiac difficulties (angina, myocardial infarction, and severe hypertension) will initially be excluded from the study due to concern that intensive EXP, often accompanied by temporary increases in heart rate and blood pressure, may pose risks of exacerbating cardiac status. They will be included once they are cleared by the cardiologist.
2. Veterans with comorbid Axis I psychotic disorders or acute substance abuse disorders initially will be excluded from the study but will be eligible once their substance abuse is under control for at least two weeks. Additionally, an Axis II diagnosis of antisocial personality disorder will be reason for exclusion.
3. Because PTSD typically is accompanied by high rates of comorbid psychiatric disorders (Keane & Wolfe, 1990), patients with comorbid depressive disorders, anxiety disorders, and personality disorders other than Antisocial Personality Disorder will be included. Also, veterans who have a diagnosis of mild Traumatic Brain Injury will be included, in order that our sample is as representative of OIF/OEF veterans as possible. We will address the issue of comorbid mTBI in the data analysis. In all cases included, PTSD must be considered the primary disorder.
4. Patients must have a symptom duration of at least 6 months.
5. Patients on benzodiazepines will be given an opportunity to discontinue and will be off benzodiazepines for at least two weeks prior to beginning the study. This exclusion is based on the empirical evidence to suggest that the efficacy of EXP for other anxiety disorders may be attenuated by benzodiazepines (Gray, 1987; Wardle, 1990). Patients on SSRI antidepressant medication for PTSD (Ballenger et al., 2000; Brady et al., 2000) will be included once their medication regimen has stabilized for at least 2 weeks. SSRI medication dosage must remain stable throughout the course of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Clinician-Administered PTSD Scale (CAPS; Blake et al., 1990; Weathers & Litz, 1994; Weathers et al., 1999) | after 17 weeks for two study arms; after three weeks for the third study arm
  PTSD Symptom Severity

SECONDARY OUTCOMES:
Quality of Life Questionnaire (QLQ; Evans & Cope, 1989) | after 17 weeks for two study arms; after three weeks for the third study arm
Clinician-Administered PTSD Scale (Selected items) | after 17 weeks for two study arms; after three weeks for the third study arm
  We will examine a subset of the CAPS separately, using frequency and intensity ratings on 4 items (interest in activities, social detachment, range of affect, anger control). These items were independently rated by 3 of the study investigators as being representative of social/emotional functioning
Objective Functional Indicators | after 17 weeks for two study arms; after three weeks for the third study arm
  Data will be collected via a clinician-administered rating form regarding objective indicators of social functioning, such as changes in marital status, employment status, residential status, legal involvement, psychiatric hospitalization, and utilization of medical care.
Clinical Global Impressions Scale | after 17 weeks for two study arms; after three weeks for the third study arm
  The Severity and Global Improvement Subscales are each 7-point scales which are part of the ECDEU Assessment Manual for Psychopharmacology. They will be used to assess overall severity and improvement. The CGI severity rating is a frequently used measure in pharmacological treatment studies and could be useful in making comparisons of rates of improvement from this study and those of drug studies.
Health-Related Functioning: Medical Outcome Study Short Form-36 Health Survey | after 17 weeks for two study arms; after three weeks for the third study arm
  The SF-36 is a 36-item questionnaire that measures health status and functioning over the past four weeks
Patient Ratings | after 17 weeks for two study arms; after three weeks for the third study arm
  For a one-week period at each assessment point, patients will keep a log of daily symptoms, such as nightmares, flashbacks, total hours of sleep, and exaggerated startle responses behavioral ratings to monitor the frequency and severity (on a 10-point scale) of PTSD
The PTSD Checklist (PCL-M; Weathers et al., 1993) | after 17 weeks for two study arms; after three weeks for the third study arm
  PTSD Symptom Severity

OTHER OUTCOMES:
Treatment Credibility | after week 3 for 17 week arms; after third day for 3 week arm
  To assess for differences in outcome expectancy, treatment credibility scales developed by Borkovec and Nau (1972) will be used. Four of the questions will be used for this study, with 10-point Likert scales. These include questions regarding how logical the treatment seems, how confident participants are about treatment, and their expectancy of success.
Charleston Psychiatric Outpatient Satisfaction Scale (CPOSS-VA; Frueh et al., 2002): | after 17 weeks for two study arms; after three weeks for the third study arm
  The CPOSS-VA is 16-item measure, with a Likert scale response format, based on a general measure of patient satisfaction (Pellegrin et al., 2001).

CONTACTS AND LOCATIONS:
Overall Officials: Deborah C Beidel, Ph.D., ABPP, Principal Investigator — University of Central Florida
Locations (1):
- University of Central Florida, Orlando, Florida, United States